CLINICAL TRIAL: NCT04793347
Title: Effect of Shock Waves Therapy on Anal Fissure
Brief Title: Effect of Shock Waves Therapy on Chronic Anal Fissure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: amr bayoumi salama (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, amr bayoumi salama, faculty of physical therapy. Cairo university, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nu5332
Record Dates: First submitted 2021-03-06; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Chronic Anal Fissure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- shock waves (Experimental): group of patients with anal fissure will be treated with shock waves
  Interventions: Device: shock master (shock waves device)

INTERVENTIONS:
Device: shock master (shock waves device) — device produces shock waves

SUMMARY:
the study conducted to assess if there is an effect of Extracorporeal Shock Wave Treatment on anal fissure

DETAILED DESCRIPTION:
Design of the study:

A prospective, randomized, blind, paired (right/left) comparison.

Materials:

Measurement tool:

* healing of anal fissure,
* Wexner Constipation Scoring System
* anal pain intensity by means of a 10-point visual analogue scale (VAS)

Therapeutic instruments:

•. shock waves

• topical application of 0.4% glyceryl trinitrate (GTN) ointment

Methods:

• Testing procedures: The assessment will be performed before commencing treatment, after 4 and 8 weeks of the treatment.

• Treatment procedures: Patients will be assigned randomly into two groups equal in number: shock waves Group: twenty patients will receive the shockwaves on perianal area of for 4 weeks (3 sessions /week). control Group: twenty patients will receive the recommended routine medical treatment include topical application of 0.4% glyceryl trinitrate (GTN) ointment only..

ELIGIBILITY:
Inclusion Criteria:

* patient with chronic anal fissure
* symptomatic for at least 6 months
* failed conservative measures

Exclusion Criteria:

* Pregnant women,
* cardiac patients,
* patients with a pacemaker,
* low molecular heparin or warfarin treatment,
* neurological disease,

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
VAS | up to 3 months
  assessment of pain

SECONDARY OUTCOMES:
wexener scale | up to 3 months
  assess the constipation

CONTACTS AND LOCATIONS:
Locations (1):
- Amr, Giza, Egypt